CLINICAL TRIAL: NCT04615143
Title: Tislelizumab or Tislelizumab Combined With Lenvatinib Neo-adjuvant Treatment for Resectable Recurrent Hepatocellular Carcinoma：Phase II Non-randomized Control Clinical Trial
Brief Title: Tislelizumab or Tislelizumab Combined With Lenvatinib Neo-adjuvant Treatment for Resectable RHCC
Acronym: TALENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHCC2020
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Hepatocellular Carcinoma
Keywords: recurrent hepatocellular carcinoma; neoadjuvant treatment; immune therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab (Experimental): Tislelizumab is one kind of PD-1 inhibitors. Patients enrolled will receive Tislelizumab as neoadjuvant treatment before surgery (200mg q3w*2 cycles) and as adjuvant treatment after surgery for 1 year
  Interventions: Drug: Tislelizumab
- Tislelizumab Combined Lenvatinib (Experimental): Patients enrolled will receive Tislelizumab combined Lenvatinibas neoadjuvant treatment before surgery (Tislelizumab: 200mg q3w*2 cycles+Lenvatinib 8/12mg qd*4weeks) and as adjuvant treatment after surgery for 1 year
  Interventions: Drug: Tislelizumab combined with Levatinib

INTERVENTIONS:
Drug: Tislelizumab — Patients receive Tislelizumab on week 1 and week 4 (200mg, iv, q3w). After 2 cycles of Tislelizumab and evaluation of resectability, patients will receive surgery in 6 weeks after enrollment. Patients will receive Tislelizumab for 1 year (200mg, iv, q3w, 17 cycles) in 4-6 weeks after surgery.
  Arms: Tislelizumab
Drug: Tislelizumab combined with Levatinib — Patients receive Tislelizumab on week 1 and week 4 (200mg, iv, q3w); Lenvatinib from Day1 to Day 28 (8/12mg qd). After neoadjuvant treatment and evaluation of resectability, patients will receive surgery in 6weeks after enrollment. Patients will receive Tislelizumab combined with Lenvatinib for 1 year in 4-6 weeks after surgery.
  Arms: Tislelizumab Combined Lenvatinib

SUMMARY:
This non-randomized phase II clinical trial aimed to explore the efficacy and safety of Tislelizumab or Tislelizumab combined with Lenvatinib as neoadjuvant treatment for resectable RHCC patients

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) patients have about 70% of 5-year recurrence rate after curative treatment. Only 30% of recurrent HCC (RHCC) patients are resectable when diagnosed. Neoadjuvant treatment may reduce tumor burden and recurrence rate after surgery for RHCC patients. Immune checkpoint inhibitors combined with or without antiangiogenic agents have already been reported effective in advanced HCC patients as first-line therapy, and in several early-stage solid tumors as neoadjuvant therapy. According to several preclinical results, immune infiltration and the expression of PD-1 were higher in RHCC tumors than in paired primary tumors. So, immune checkpoint inhibitors combined with or without antiangiogenic agents might have a better response in RHCC patients than primary HCC patients. Herein, we designed this phase II clinical trial to explore the efficacy and safety of Tislelizumab (PD-1 inhibitor) or Tislelizumab combined with Lenvatinib as neoadjuvant treatment for resectable RHCC patients. Enrolled resectable RHCC patients will be divided into two non-randomized seperate arms, sequentially (arm 1: neoadjuvant tislelizumab; arm 2: neoadjuvant tislelizumab and lenvatinib). Each arm was estimated to enroll 40 patients. We have already enrolled 17 patients in arm 1, and have terminated the enrollment of arm 1 due to modest treatment responses. The enrollment of arm 2 is ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as recurrent hepatocellular carcinoma after curative treatment;
2. The criteria for resectability is met;
3. Has at least one evaluable lesion according to the RECIST 1.1 standard and has not received local treatment;
4. Eastern Cooperative Oncology Group score 0-1, Child-pugh score 5-7;
5. Agree to biopsy and blood sample collection;
6. Adequate organ and marrow function.

Exclusion Criteria:

1. Previously received any transarterial chemoembolization and immune therapy and other local or systemic liver cancer treatments, except for curative ablation;
2. Extrahepatic metastasis;
3. History of gastroesophageal varices or active cardia ulcers associated with a high risk of bleeding;
4. History of autoimmune disease or need to take immunosuppressant drugs for a long time;
5. History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
6. Abnormal organ function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate | 1 year
  Defined as the percent of patients without recurrence, progression or death in one year after enrollment

SECONDARY OUTCOMES:
Objective response rate | At time of surgery
  Defined as the percent of patients with a complete response (CR) or partial response (PR) documented by the Investigator per RECIST 1.1.
Incidence of severe adverse events | Three months after treatment
  Defined as the percent of patients with adverse events over grade 3.
Major pathological response rate | At time of surgery
  Defined as the percent of patients with less than 10% visible cancer cells out of the surface expression of the total tumor area at the time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No